CLINICAL TRIAL: NCT00094419
Title: The Role of Complementary and Alternative Medicine (CAM), Folk Care and Faith-Based Approaches in the Home Management of Persistent Asthma in Low-Income African American and Caucasian Adults
Brief Title: Complementary and Alternative Medicine Use in Low-Income African American and Caucasian Adults With Asthma
Status: Completed | Type: Observational
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Maureen George, Principal Investigator, Johns Hopkins School of Nursing
Other Study IDs: F32AT002012-01 (NIH)
Record Dates: First submitted 2004-10-18; First posted 2004-10-19 (Estimated); Last update posted 2008-08-12 (Estimated); Status verified 2008-08

CONDITIONS: Asthma
Keywords: Complementary Therapies
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to identify the types of and frequency of use of complementary and alternative medicine (CAM) strategies among low-income Caucasian and African American adults with persistent asthma. The overall goal is to collect data that will increase understanding of health beliefs and behaviors in people with low-income backgrounds so that studies can be created that may help modify and improve patients' symptoms of asthma.

DETAILED DESCRIPTION:
The rates of asthma-related deaths and disease are disproportionately high among African Americans compared to Caucasians. Surveys indicate that middle- and upper-income Caucasians use more CAM than African Americans, but the therapies utilized are different. This study will determine how well people with persistent asthma adhere to their treatment and whether the type and frequency of use of CAM affects treatment adherence.

Participants will begin this study by taking part in an interview about adherence to their current inhaled corticosteroids (ICS) regimen and their personal CAM use. After completing the interview, participant adherence to their ICS regimen will be monitored for 6 weeks. Depending on the type of ICS participants are taking, monitoring will be conducted either by participant self-reporting or electronic monitors that record the time and date of medication inhalation. Participant adherence will also be assessed at study completion.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed asthma with episodes that last for long periods of time
* Medicaid recipients
* Self-identify as African American or Caucasian
* Daily use of inhaled corticosteroids
* Able to speak English
* Have mental capacity to understand and participate in the study

Exclusion Criteria:

* Prisoners
* History of smoking at least ten packs of cigarettes per year
* Currently smoke more than one and a half packs of cigarettes per week

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2004-11; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen George, PhD RN AE-C, Principal Investigator — Johns Hopkins Medical Institute
Locations (2):
- United States (2):
  - Johns Hopkins Bayview Campus, Baltimore, Maryland
  - Presbyterian Medical Center at the University of Pennsylvania, Philadelphia, Pennsylvania